CLINICAL TRIAL: NCT00439543
Title: Inhaled Iloprost in Pulmonary Hypertension Secondary to Pulmonary Fibrosis
Brief Title: Trial of Iloprost in Pulmonary Hypertension Secondary to Pulmonary Fibrosis
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Interstitial Lung Disease Study Group, Korea (Network)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TILOPF
Record Dates: First submitted 2007-02-22; First posted 2007-02-23 (Estimated); Last update posted 2007-02-23 (Estimated); Status verified 2007-02

CONDITIONS: Pulmonary Fibrosis; Pulmonary Hypertension
Keywords: Pulmonary fibrosis; pulmonary hypertension; Iloprost; Efficacy
MeSH Terms: conditions — Pulmonary Fibrosis; Hypertension, Pulmonary

INTERVENTIONS:
Drug: Iloprost inhalation

SUMMARY:
Idiopathic pulmonary fibrosis(IPF) is chronic progressive fibrosing lung disease of unknown cause. There is no effective therapy yet for this disease and the mean survival in most reports is about 3 years after the diagnosis. Because of the stiff fibrosis of the lung, pulmonary hypertension is the late complication of IPF and its development heralds a very poor outcome of the patients. For the primary pulmonary hypertension, recently the effective drugs have been available. However, there is no study about the efficacy of these drugs in the patients with pulmonary hypertension secondary to pulmnary fibrosis, and the aim of this trial is to study the safty and efficacy of "Iloprost," one of the safe and effective drugs in primary pulmonary hypertension.

DETAILED DESCRIPTION:
* Prospective open labeled observational study
* Subjects: About 15 patients with secondary pulmonary hypertension due to IPF or pulmonary fibrosis associated with collagen vascular diseases.
* Method: 3 month trial of inhaled iloprost. Check the safty and measure the pulmonary arterial pressure by right heart catheterization, exercise capacity by 6 minute walking test, echocardiography, and quality of life questionnaires before and after the trial.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of idiopathic pulmonary fibrosis or fibrotic NSIP according to American Thoracic Society and European Respiratory Society guidelines by biopsy and diagnosis of pulmonary fibrosis associated with connective tissue disease.
* Mean pulmonary artery pressure over 30mmHg.
* NYHA functional class II to IV

Exclusion Criteria:

* Suffering lung diseases other than pulmonary fibrosis (COPD, Pulmonary Thromboendarterectomy ).
* Administration of prostanoids, bosentan, beta- blocker or phosphodiesterase5 inhibitor.
* Dosage adjustment of calcium channel blockers within 6 weeks.
* Resting pulmonary capillary wedge pressure over 15mmHg.
* Bleeding tendency.
* Bilirubin level above 3mg/dl or creatinine clearance level below 30ml/min.
* Unstable angina pectoris, myocardial infarction or severe arrhythmia within 6 months.
* Cerebrovascular accident within 6 months.
* Present lung infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15
Dates: Start 2007-03; Study Completion 2007-08

PRIMARY OUTCOMES:
Safety
Pulmonary arterial pressure
Exercise capacity (6 minute walking test)

SECONDARY OUTCOMES:
6 minute walking test: Min. oxygen saturation.
NYHA class,
Quality of life (St. George Respiratory questionnaires)
Pulmonary vascular resistance, cardiac output.
Increment of pulmonary arterial pressure after the exercise
6) Pulmonary function test

CONTACTS AND LOCATIONS:
Overall Officials: Dong Soon Kim, MD, Principal Investigator — Asan Medical Center, Ulsan University, Seoul, Korea, Republic of
Locations (1):
- Pulmonary Medicine, Asan Medical Center, Ulsan University, Seoul, South Korea